CLINICAL TRIAL: NCT00866502
Title: A Randomized, Double-blind, Placebo Controlled, Safety and Tolerability Study of Intracerebroventricular Administration of sNN0031 to Patients With Idiopathic Parkinson's Disease (PD) of Moderate Severity, Using an Implanted Catheter and a SynchroMed® II Pump.
Brief Title: A Safety and Tolerability Study of Intracerebroventricular Administration of sNN0031 to Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Newron Sweden AB (Industry)
Collaborators: Medtronic (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sNN0031-001; Q-26239
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; Safety; PDGF; Intracerebroventricular; Infusion; Device
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sNN0031 (Experimental): Continuous ICV infusion for two weeks at one of three dose levels
  Interventions: Drug: sNN0031
- Placebo (Placebo Comparator): Continuous ICV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sNN0031 — Continuous ICV infusion for two weeks
  Other Names: PDGF
  Arms: sNN0031
Drug: Placebo — Continous ICV infusion
  Other Names: Artificial CSF
  Arms: Placebo

SUMMARY:
This study is conducted to evaluate the safety and tolerability of the drug product sNN0031, containing Platelet Derived Growth Factor (PDGF), when administered directly into one of the fluid filled cavities in the brain using an implanted catheter and an implanted SynchroMed® II pump. Patients with a diagnosis of Parkinson's disease will be enrolled.

DETAILED DESCRIPTION:
Tremor, rigidity, slow movement, poor balance, and difficulty walking are characteristic symptoms of Parkinson's disease (PD) that are associated with degeneration of dopamine-producing nerve cells in the brain. Administration of growth factors that stimulate neuronal stem and progenitor cells is one possible approach to restore the dopaminergic activity. The drug product sNN0031 containing the endogenous growth factor PDGF has been demonstrated to reduce the typical symptoms in animal models of PD.

NeuroNova intends to investigate whether intracerebroventricular administration of PDGF in the form of the drug product sNN0031 can improve motor function in patients with PD. In this first study the safety and tolerability of treatment for 2 weeks followed by 10 weeks follow-up will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. Females should either be post-menopausal (at least 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with FSH levels >40 mIU/mL), be surgically sterilized (bilateral oophorectomy w/o hysterectomy), or use adequate contraception (oral contraceptives, intrauterine device or double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam.) during the duration of the study.
* Diagnosis of idiopathic Parkinson's disease (PD) of moderate severity (modified Hoehn & Yahr Stage IIb-III).
* Effect duration of oral L-dopa dose intake ≤4 hours
* Score ≥30 on motor part (part III) of UPDRS at defined off (>12 hours after last dose intake)
* Dopaminergic responsiveness with at least 33% decrease in the UPDRS part III score after administration of L-dopa
* Disease duration at least 5 years
* Age 30 to 75 years
* Stable anti-Parkinson treatment for at least 3 months
* Ophthalmologic examination with normal findings regarding vascular structure and function
* MRI examination of the brain and cervical spinal cord within 3 months before anticipated implantation of the device with no findings of tumors or potential sources of pathological bleedings, or abnormality that may interfere with the assessments of safety or efficacy or would, in the judgment of the investigator, represent a surgical risk to the subject.
* Values of coagulation parameters including platelet count, normalized prothrombin complex (PK-INR), activated partial thromboplastin time (APTT) within normal ranges.
* The subject is medically able to undergo the surgery required for stereotactic implantation of the catheter and infusion pump.
* Has been given written and verbal information, has had opportunity to ask questions about the study, and understands time and procedural commitments
* Signed consent (written) to participate in the study

Exclusion Criteria:

* Atypical form of PD including repeated head trauma, drug- or toxin-induced PD, and other neurological conditions including Shy-Drager syndrome (multiple system atrophy), progressive supranuclear palsy, Wilson's disease, Huntington's disease, Hallervorden-Spatz syndrome, Alzheimer's disease, Creutzfeldt-Jakob disease, olivopontocerebellar atrophy, and post-traumatic encephalopathy
* Concurrent dementia with a score of 20 or lower on the MMT rating scale
* Concurrent clinically significant depression with a score of 16 or higher on the MADRS rating scale, equivalent to moderate or severe depression.
* Exposure to neuroleptic drugs blocking dopamine receptors within 6 months
* History of structural brain disease including tumors and hyperplasia
* History of increased intracranial pressure
* Prior surgical procedures or implantation of device for the treatment of PD
* Prior exposure to any formulation of PDGF-BB (including topical)
* Uncontrolled hypertension with blood pressure >160 mmHg systolic or >90 mmHg diastolic.
* Any disorder that precludes a surgical procedure (eg, signs of sepsis or inadequately treated infection), alters wound healing (e.g. including bleeding disorders), or renders chronic ICV delivery or device implants medically unsuitable.
* Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that is not managed optimally. Physicians should specifically investigate anatomical factors at or near the implant site (e.g., vascular abnormalities, neoplasms, or other abnormalities), underlying disorders of the coagulation cascade, platelet function, or platelet count (e.g., hemophilia, Von Willebrand's disease, liver disease, or other medical conditions), and the administration of any antiplatelet or anticoagulant medication (e.g., aspirin, Plavix, NSAIDs) in the pre- or perioperative period. Any of those conditions or drugs could place a patient at an increased risk for intraoperative or postoperative bleeding.
* Presence of an implanted shunt for the drainage of cerebrospinal fluid (CSF) or an implanted central nervous system (CNS) catheter.
* Presence of cardiac pacemakers, spinal cord stimulators, implantable programmable intraspinal drug pumps, or any other device that may interfere or interact with the programmer, without prior approval by Medtronic.
* Clinically significant abnormalities in hematology or clinical chemistry parameters as assessed by the investigator
* Ongoing medical condition that according to the investigator would interfere with the conduct and assessments in the study. Examples are medical disability (eg, severe degenerative arthritis, compromised nutritional state, peripheral neuropathy) that would interfere with the assessment of safety and efficacy of investigational product or device performance, or would compromise the ability of the subject to undergo study procedures (eg, MRI, PET), or to give informed consent.
* Participation in another clinical trial with an investigational drug or device within 3 months prior to Screening visit.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability through assessment of adverse events, ECGs, vital signs, clinical laboratory variables, MRI of brain and spinal cord, CSF sampling, and device performance as characterized by catheter tip placement and infusion accuracy. | Multiple over 3 months

SECONDARY OUTCOMES:
Time course of PD disease activity as measured by the UPDRS, MADRS and MMT rating scales. | Multiple over 3 months
Change in caudate and putamen dopamine turnover using PET scans of 11C-PE2I uptake | Baseline and at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sven Pålhagen, MD, Principal Investigator — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Huddinge, Stockholm

REFERENCES:
- [Derived] Paul G, Zachrisson O, Varrone A, Almqvist P, Jerling M, Lind G, Rehncrona S, Linderoth B, Bjartmarz H, Shafer LL, Coffey R, Svensson M, Mercer KJ, Forsberg A, Halldin C, Svenningsson P, Widner H, Frisen J, Palhagen S, Haegerstrand A. Safety and tolerability of intracerebroventricular PDGF-BB in Parkinson's disease patients. J Clin Invest. 2015 Mar 2;125(3):1339-46. doi: 10.1172/JCI79635. Epub 2015 Feb 17. PMID 25689258